CLINICAL TRIAL: NCT01081379
Title: The Relation Between the Maternal Cellular Immune System and Cytomegalovirus Intrauterine Infection
Brief Title: The Maternal Cellular Immune System and Cytomegalovirus Intrauterine Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Yedidia Yifat, Yechiel Schlesinger, MD, Shaare Zedek Medical Center., Shaare Zedek Medical Center
Other Study IDs: Schlesinger - CMV
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Pregnant Women; Cytomegalovirus Infections
Keywords: Cytomegalovirus Infections; Pregnancy; T-Lymphocytes; Transmission
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pre-conception immunity: pre-conception immunity- pregnant women with CMV seropositive
- primary CMV infection: primary CMV infection- pregnant women with primary CMV infection (defined as CMV IgG sero-conversion, the presence of low avidity IgG antibodies or the presence of IgM with no previous IgG antibodies).

SUMMARY:
The purpose of this study is to find a correlation between function of cytomegalovirus -specific T cells and the probability for intrauterine transmission.

DETAILED DESCRIPTION:
Fetal infection with CMV is the most common cause of intrauterine infection. Only 40% of pregnant women with primary CMV transmit the virus to their fetus. Many of these women are referred to amniocentesis and many elect to terminate pregnancy without knowledge about fetal infection or damage. Currently it is assumed that transmission is dictated by variety of factors including maternal and fetal immune system. Efforts to find correlation between maternal immune system and fetal infection which can be used as a diagnostic marker were unsuccessful.

Our hypothesis is that there is a correlation between cellular immune response of the mother to CMV infection and viral transmission to the fetus.

Pregnant women with primary CMV infection (40% of whom are expected to be transmitters)and with pre-conception immunity will participate in this study.

Blood from these women will be incubated with CMV peptides and T cell activation will be measured by the secretion of various cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* CMV IgG sero-conversion or the presence of low avidity IgG antibodies or the presence of IgM with no previous IgG antibodies.

Exclusion Criteria:

* Underlying immune deficiencies
* Other pregnancy complications

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women with primary CMV
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Maternal-Fetal transmission of CMV | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yechiel Schlesinger, M.D., Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel